CLINICAL TRIAL: NCT00326092
Title: A Study of a Glaucoma Therapy to Treat Open-Angle Glaucoma or Ocular Hypertension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C-05-49
Record Dates: First submitted 2006-05-12; First posted 2006-05-16 (Estimated); Last update posted 2016-11-18 (Estimated); Status verified 2007-09

CONDITIONS: Open-angle Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — brinzolamide; Timolol

INTERVENTIONS:
Drug: Brinzolamide/Timolol

SUMMARY:
The purpose of this study is to assess the comfort of a glaucoma therapy in patients with open-angle glaucoma or ocular hypertension

ELIGIBILITY:
Inclusion Criteria:

* Adults of either sex and any race diagnosed with open-angle glaucoma (with or without pseudoexfoliation or pigment dispersion component)

Exclusion Criteria:

* Under 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88
Dates: Start 2006-05; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Ocular discomfort

CONTACTS AND LOCATIONS:
Overall Officials: Julia White, Study Director — Study Director
Locations (1):
- Fort Worth and Other Sites, Fort Worth, Texas, United States

REFERENCES:
- [Result] Vold SD, Evans RM, Stewart RH, Walters T, Mallick S. A one-week comfort study of BID-dosed brinzolamide 1%/timolol 0.5% ophthalmic suspension fixed combination compared to BID-dosed dorzolamide 2%/timolol 0.5% ophthalmic solution in patients with open-angle glaucoma or ocular hypertension. J Ocul Pharmacol Ther. 2008 Dec;24(6):601-5. doi: 10.1089/jop.2008.0030. PMID 19049301